CLINICAL TRIAL: NCT06936449
Title: Long-term Follow-up of a Cohort of Adult CI632D and CI632 Participants in the CLTD5759 CI-DEX Study
Brief Title: Long-term Follow-up of a Cochlear Implant With Dexamethasone Eluting Electrode Array
Acronym: CI-DEX-LTFU
Status: Recruiting | Type: Observational
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Other Study IDs: CLTD5759-S1
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-05

CONDITIONS: Sensorineural Hearing Loss; Bilateral Hearing Loss
Keywords: cochlear implant; dexamethasone; bilateral hearing loss; sensorineural hearing loss
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss, Bilateral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: CI632D Investigational Medical Device (IMD): Adults with bilateral postlinguistic sensorineural hearing loss, who have received the CI632D cochlear implant
  Interventions: Device: CI632D
- Active Comparator: CI632 Comparator Device: Adults with bilateral postlinguistic sensorineural hearing loss, who have received the CI632 cochlear implant
  Interventions: Device: CI632

INTERVENTIONS:
Device: CI632D — CI632 cochlear implant with Slim Modiolar electrode including dexamethasone in the electrode within wells
  Groups: Experimental: CI632D Investigational Medical Device (IMD)
Device: CI632 — CI632 cochlear implant with Slim Modiolar electrode with market approval and does not include dexamethasone
  Groups: Active Comparator: CI632 Comparator Device

SUMMARY:
A long-term follow-up of Cochlear's cochlear implant electrode array which passively elutes dexamethasone for a defined period of time to help reduce inflammatory responses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed study obligations of the CLTD5759 CI-DEX study and enrolled at a site selected for participation.
* Subjects implanted with a CI632D or a CI632 cochlear implant under the CLTD5759 (NCT04750642).
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Unrealistic expectations on the part of the subject, regarding the possible benefits, risks, and limitations that are inherent to participation as determined by the Investigator.
* Additional disabilities that may affect the subject's participation or safety during the clinical investigation.
* Unable or unwilling to comply with all the requirements of the clinical investigation as determined by the Investigator.
* Currently participating, or participated within the last 30 days, in another interventional clinical investigation/trial involving an investigational drug or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals available from those sites invited to participate in the study consisting of up to 10 subjects implanted with the CI632D and up to 9 subjects with the CI632 in the CIDEX study (NCT04750642)
Sampling Method: Non-Probability Sample
Enrollment: 19 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Comparison of Monopolar (MP1+2) Impedance Measurement (kOhms) between groups obtained in the CLTD5759 (NCT04750642) study, and at the 2 through 5 years post-activation routine follow-up visits. | 5 years post-activation

SECONDARY OUTCOMES:
Comparison of CI632D and CI632 device-related adverse events between groups from enrolment in this study through 5 years postactivation. | 5 years post-activation
Comparison of Four-point Impedance Measurement between groups obtained in the CLTD5759 (NCT04750642) study, and from enrolment in this study through 5 years postactivation. | 5 years post-activation
Comparison of low-frequency acoustic hearing between groups as measured by pure tone average thresholds over the range 125 through 500 Hz, obtained in the CLTD5759 (NCT04750642) study and from enrolment in this study through 5 years postactivation. | 5 years post-activation
Comparison of speech perception in quiet (CNC word scores) for the best unilateral listening condition in the implanted ear between groups obtained in the CLTD5759 (NCT04750642) study, and from enrolment in this study through 5 years postactivation. | 5 years post-activation
Speech perception in noise (AzBio sentence scores) for the best bilateral listening condition obtained between groups in the CLTD5759 (NCT04750642) study, and from enrolment in this study through 5 years postactivation. | 5 years post-activation

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Rocky Mountain Ear Center, Englewood, Colorado
  - University of Iowa, Iowa City, Iowa
  - University Hospitals Cleveland, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No